CLINICAL TRIAL: NCT01430507
Title: A Phase IIb, 12 Week Randomized, Double-Blind, Parallel Group, Placebo-Controlled Study to Evaluate Efficacy, Safety and Tolerability of Revamilast in Patients With Active Rheumatoid Arthritis Who Have Had an Inadequate Response to Methotrexate
Brief Title: A Clinical Trial to Study the Effects of Revamilast in Patients With Rheumatoid Arthritis
Acronym: TERRA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Glenmark Pharmaceuticals Ltd. India (Industry)
Collaborators: Glenmark Pharmaceuticals S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GRC 4039-203; 2011-000107-40 (EudraCT Number)
Record Dates: First submitted 2011-09-07; First posted 2011-09-08 (Estimated); Last update posted 2012-12-28 (Estimated); Status verified 2012-08

CONDITIONS: Rheumatoid Arthritis
Keywords: Anti-inflammatory drugs, DMARD
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Medium Dose (Experimental): Medium Dose Revamilast
  Interventions: Drug: Revamilast
- High Dose (Experimental): High Dose Revamilast
  Interventions: Drug: Revamilast
- Placebo (Placebo Comparator): Matching Placebo in Triple Dummy Format
  Interventions: Drug: Placebo Comparator
- Low dose (Experimental): Low dose Revamilast
  Interventions: Drug: Revamilast

INTERVENTIONS:
Drug: Revamilast — Tablet, Low dose, Once daily for 12 weeks
  Arms: Low dose
Drug: Revamilast — Tablet, Medium dose, Once daily for 12 weeks
  Arms: Medium Dose
Drug: Revamilast — Tablet, High dose, Once daily for 12 weeks
  Arms: High Dose
Drug: Placebo Comparator — Matching Placebo in triple dummy format, Tablet, Once daily for 12 weeks
  Arms: Placebo

SUMMARY:
Rheumatoid arthritis (RA) is a systemic autoimmune and chronic inflammatory disease that causes progressive damage to joints of the body, affecting the functional capacity. Effective management of patients with RA requires a multidisciplinary approach. Despite the various combinations, there is a significant population of RA patients who are not responding to these combinations or showing inadequate response to methotrexate alone. Hence, there is a need for a unique combination of drugs targeting different pathological process to yield the best results in those patients where prognosis is poor. Combination of revamilast with first line therapy like methotrexate could provide better treatment options to a larger population of RA patients having moderate to severe disease and who are inadequately controlled on one or the other DMARDs.

This is randomized, double-blind, placebo-controlled, parallel group study. The study will include patients with active RA receiving stable and maximum tolerated dose of MTX.

Patients will be recruited after providing written informed consent. After screening and run in period (single blind placebo for 4 weeks), patients will be randomized (meeting randomization criteria) in 1:2:2:2 ratios to receive either one of three doses (Low, Medium and High) of revamilast or placebo along with MTX.

The primary objective of the study is to determine the percentage of patients achieving ACR20 response at 12 weeks. Secondary objectives include determining percentage of patients with ACR50 and ACR70 response, change in DAS-28 score, change in serum CRP and ESR values and frequency and use of rescue medication.

During the treatment period, there will be 5 further study visits at week 2, week 4, week 8, week 12, for efficacy, safety and tolerability assessment and visit at week 14 will be follow up visit.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 to ≤ 65 years of age
2. Documented history of RA; diagnosed according to the revised American College of Rheumatology criteria (ACR)
3. Active RA defined as patients with:

   * 6 swollen joint counts
   * 6 tender/painful joint counts, and

     * At least two of the three following criteria:

       * Rheumatoid Factor positive or Anti CCP positive
       * CRP ≥1.2 times upper limit of normal reference range or ESR >28 mm/hr
       * Morning stiffness lasting >45 min for at least last4 weeks
4. DAS-28 CRP values ≥ 4.5 at screening (visit 1)
5. Patients must have been on stable (15 mg to 25 mg) or maximum tolerated dose of MTX for at least 12 weeks prior to screening
6. The patient's written informed consent to participate in the study
7. Female participants must have a negative serum pregnancy test at screening visit.
8. Males must agree to use barrier while on study medication and for 90 days after taking the last dose of study medication
9. Must meet the following laboratory criteria:

   * Hemoglobin ≥ 9 g/dL
   * White blood cell (WBC) count; ≥3.0 X 109/L
   * Platelet count ≥ 100,000 /L (100 X 109/L)
   * Serum creatinine <1.5 mg/dL (or 133mol/L)
   * Total bilirubin <2.0 mg/dL
   * AST & ALT<1.5 times upper limit of normal

Exclusion Criteria:

1. Diagnosis of RA prior to 16 years of age (Juvenile RA)
2. Non-degenerative joint diseases or other joint diseases that could interfere with the evaluation of RA
3. Patients with any other autoimmune rheumatic disorders with the exception of Sjogren's syndrome.
4. Patients with first degree relative with immune deficiency
5. History of infection with human immunodeficiency virus and/or active hepatitis B or C
6. Severe disabling arthritis leaving the patient eligible for surgical intervention, or incapacitated and prostrated patients
7. Patients with a history of drug or alcohol abuse or chronic smoking
8. Uncontrolled diabetes mellitus
9. Concurrent diseases that might interfere with the conduct of the study,
10. ECG abnormalities judged by the investigator to be clinically significant
11. History of using any other test drug, one month before the beginning of this trial
12. Women who are pregnant or breast-feeding or on hormonal therapy
13. Patients who in the Investigator's opinion might not be suitable for the study.
14. Patients with a life expectancy of less than 1 year

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2011-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Percentage of patients achieving ACR20 response | 12 weeks

SECONDARY OUTCOMES:
Percentage of patients achieving ACR50 and ACR 70 response | 12 weeks
Change in DAS-28 score | week 12
Change in serum CRP and ESR values | 12 weeks
Frequency and use of rescue medication | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dr Lalit Lakhwani, Study Director — Glenmark Pharamceuticals SA
Locations (36):
- India (16):
  - Advance Rheumatology Clinic, Hyderabad, Andhra Pradesh
  - Mahavir Hospital and Research Center, Hyderabad, Andhra Pradesh
  - Sri Deepti Rheumatology Center, Hyderabad, Andhra Pradesh
  - Krishna Institute of Medical Sciences, Secunderabad, Andhra Pradesh
  - Rathi Orthopaedic & Research Center, Ahmedabad, Gujarat
  - Shalby Hospitals, Ahmedabad, Gujarat
  - Centre for Knee & Hip Surgery, Vadodara, Gujarat
  - Chanre Rheumatology and Immunology centre and Research, Bangalore, Karnataka
  - M S Ramaiah Medical College and Hospital, Bangalore, Karnataka
  - Kennisha Rheumatology Care & Diagnostics, Mumbai, Maharashtra
  - Sushrut Hospital Research Centre and PG Institute of Orthopaedics, Nagpur, Maharashtra
  - Vidarbha Arthritis & Superspeciality Clinic, Nagpur, Maharashtra
  - Chennai Meenakshi Multispeciality Hospital Limited, Chennai, Tamil Nadu
  - Chhatrapati Shahuji Maharaj Medical University, Lucknow, Uttar Pradesh
  - Sanjay Gandhi Postgraduate Institute of Medical Sciences, Lucknow, Uttar Pradesh
  - Institute of Post Graduate Medical Education & Research (IPGMER), Kolkata, West Bengal
- Philippines (7):
  - Internal Medicine and Rheumatology, Chong Hua Hospital, Cebu, Cebu
  - Brokenshire Memorial Hospital, Davao City, Davao Region
  - Department of Medicine, Davao Doctor's Hospital, Davao City, Davao Region
  - University of Perpetual Help Dalta Medical Center, Las Piñas, National Capital Region
  - Manila Doctors Hospital, Manila, National Capital Region
  - University of Santo Tomas Hospital, Manila, National Capital Region
  - St. Luke's Medical Center, Quezon City, National Capital Region
- Poland (7):
  - Oddział Kliniczny Reumatologii i Ukladowych Chorob Tkanki Lacznej, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - NZOZ Reumed, Lublin, Lublin Voivodeship
  - Osrodek Badan Klinicznych Prof. Dr hab. med., Lublin, Lublin Voivodeship
  - Niepubliczny Zaklad Opieki Zdrowotnej Medica Pro Familia Sp. z o.o., Warszawa, Lublin Voivodeship
  - Centrum Medyczne MEDENS S.C. Grupowa Praktyka Lekarska, Chełm Śląski, Silesian Voivodeship
  - Specjalistyczna Praktyka Lekarska Joanna Badowska, Częstochowa, Silesian Voivodeship
  - Wojewodzki Zespol Specjalistycznej Opieki Zdrowotnej, Wroclaw, Silesian Voivodeship
- Sri Lanka (4):
  - Colombo South Teaching Hospital, Colombo, Colombo
  - National Hospital of Sri Lnka, Colombo, Colombo
  - Nawaloka Hospitals PLC, Colombo, Colombo
  - Teaching Hospital Karapitiya, Galle, Colombo
- United Kingdom (2):
  - Queen's Hospital, Romford, Essex
  - The Leeds Teaching Hosptial NHS Trust, Chapel Allerton Hospital, Leeds, Yorkshire